CLINICAL TRIAL: NCT07189962
Title: A Pharmacokinetic Study of SHR8554 Injection in Chinese Patients With Renal Insufficiency and Healthy Subjects
Brief Title: A Pharmacokinetic Study of SHR8554 Injection in the Population With Renal Insufficiency and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR8554-106
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Moderate to Severe Postoperative Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal renal function group (Experimental)
  Interventions: Drug: SHR8554 Injection
- Severe renal dysfunction group (Experimental)
  Interventions: Drug: SHR8554 Injection

INTERVENTIONS:
Drug: SHR8554 Injection — SHR8554 injection.

SUMMARY:
The study is being conducted to evaluate the safety and pharmacokinetic characteristics of SHR8554 injection in subjects with renal insufficiency and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. The estimated glomerular filtration rate (eGFR) of subjects in groups must meet the corresponding standards;
3. Male or female;
4. with a body mass index (BMI) between 18.0 and 28.0 kg/m2.

Exclusion Criteria:

1. History of clinically significant allergies, known allergy to SHR8554, or any other structural analogs;
2. Subjects with positive tests for infectious diseases;
3. Pregnancy or lactation women, or a fertility male or female is not willing to contraception during test;
4. Unable to tolerate venipunctures or have a history of fainting needles and blood;
5. Historic abuse of alcoholic beverages;
6. Smoke ≥ 10 cigarettes per day within 3 months prior to the study;
7. History of drug abuse;
8. Diseases with abnormal clinical manifestations that occurred before screening or are currently occurring and need to be excluded for normal renal function group;
9. Vital signs, physical examination, 12-lead electrocardiogram, or laboratory examination deemed clinically significant by the investigator for normal renal function group;
10. History of renal transplantation and/or requirement for renal dialysis treatment during the study period for severe renal function group;
11. Urinary incontinence or anuria (e.g., < 100 mL/day) for severe renal function group;
12. Other reasons that the investigator consider it inappropriate to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of SHR8554 (Cmax). | 0 hour to 48 hours after administration.
Area under the serum concentration time curve (AUC) of SHR8554. | 0 hour to 48 hours after administration.
Half-life (t1/2) of SHR8554. | 0 hour to 48 hours after administration.
Clearance (CL) of SHR8554. | 0 hour to 48 hours after administration.
Volume of distribution (Vz) of SHR8554. | 0 hour to 48 hours after administration.

SECONDARY OUTCOMES:
Cumulative excretion (Ae) of SHR8554. | 0 hour to 48 hours after administration.
Urinary excretion fraction (fe) of SHR8554. | 0 hour to 48 hours after administration.
Renal clearance (CLr) of SHR8554. | 0 hour to 48 hours after administration.
Plasma protein binding rate of SHR8554 in patients with renal insufficiency. | 0 hour to 48 hours after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided